CLINICAL TRIAL: NCT02269774
Title: Electroanatomic Origin of Premature Atrial Beats in Patients With Paroxysmal Atrial Fibrillation Induced by Intra-thoracic Pressure Swings Simulating Obstructive Sleep Apnea
Brief Title: Origin of Premature Atrial Beats Induced by Simulated Obstructive Sleep Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the strict in- and exclusion criteria only few patients could be enrolled into the study.
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Malcolm Kohler, Malcolm Kohler, Prof MD, University of Zurich
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEK-ZH-Nr. 2014-0203
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Atrial Fibrillation; Sleep Apnea, Obstructive; Atrial Premature Complexes
Keywords: Atrial Fibrillation; Obstructive Sleep Apnea; Atrial Premature Complexes; Pulmonary Vein Isolation; Mueller Manoeuvre
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive; Atrial Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary vein isolation (Other): Intra-thoracic pressure swings induced by breathing manoeuvres during standard catheter-ablation procedure. Catheter-based electrical mapping and pressure in the left atrium and pulmonary veins during standard catheter-ablation procedure. Only patients with an apnea-hypopnea index > 5/h and documented premature atrial beats during the Mueller manoeuvre will be eligible for the catheter-based electrical mapping. Follow-up after 1 year for atrial fibrillation recurrence.
  Interventions: Procedure: Standard pulmonary vein isolation
- No intevention (No Intervention): Intra-thoracic pressure swings induced by breathing manoeuvres during ECG-monitoring. Only patients with an apnea-hypopnea index < 5/h and no premature atrial beats during the Mueller manoeuvre will be assigned to the no intervention arm.

INTERVENTIONS:
Procedure: Standard pulmonary vein isolation — The MM will be carried out during a elective standard pulmonary vein isolation procedure. The MM will be performed using an occluded mouthpiece with a small air leak to prevent complete closure of the glottis during inspiration and thus assure negative pressure throughout the entire airway. After expiration, inspiration with a target negative intrathoracic pressure of -40mmHg will be carried out against the mouthpiece.
  Arms: Pulmonary vein isolation

SUMMARY:
There is accumulating evidence for obstructive sleep apnea (OSA) as an independent risk factor for paroxysmal atrial fibrillation and for high recurrence rates of atrial fibrillation after ablation therapy. We have previously shown that simulated OSA triggers premature atrial beats (PABs) by acute changes in intra-thoracic pressure. Most episodes of atrial fibrillation are initiated by PABs. However, the origin of PABs induced by intra-thoracic pressure swings is unknown. This study investigates the origin of premature atrial beats induced by intra-thoracic pressure changes that simulate obstructive sleep apnea in patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* History of ECG-documented paroxysmal atrial fibrillation within the last 12 months and currently in sinus rhythm
* Scheduled for circumferential pulmonary venous isolation treatment
* 18 to 75 years of age
* Signed informed consent

Exclusion Criteria:

* Treated with class III anti-arrhythmic agents (at the moment of pulmonary venous isolation)
* Treated for obstructive sleep apnea
* Previous catheter ablation in the pulmonary veins or left atrium
* Severe structural heart disease
* Mental or physical disability precluding informed consent or compliance with the protocol
* Enrolled in another study that would confound the results of this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Electroanatomical origin of premature atrial beats | Participants will be followed for the duration of pulmonary vein isolation, an expected average of 3 hours
  (Loop-)Catheter-based origin detection in patients with apnea-hypopnea index > 5/h in home sleep study and documented premature atrial beats during three time points: baseline (normal breathing), inspiration through a threshold load device, and the Mueller Manoeuvre (MM). Origins will be quantitatively marked at a left atrial map.

SECONDARY OUTCOMES:
Catheter-based pressure in the left atrium and pulmonary veins during intra-thoracic pressure changes | Participants will be followed for the duration of pulmonary vein isolation, an expected average of 3 hours
  Catheter-based left atrial pressure measurement in patients with apnea-hypopnea index > 5/h in home sleep study and documented premature atrial beats during three time points: baseline (normal breathing), inspiration through a threshold load device, and the Mueller Manoeuvre. Changes in left atrial pressure will be recorded in cmH2O.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, MD, Prof, Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland